CLINICAL TRIAL: NCT06331130
Title: CT Detected Tumour Infiltration Patterns of the Mesentery in High Grade Ovarian Carcinoma (HGSOC) Patients, Their Role in Treatment Planning and Outcome Prediction and How Machine Learning Can be Applied to Identify Them.
Brief Title: Mesenteric Infiltration in Ovarian Cancer
Acronym: MIO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Danube University Krems (Other); Institut du Cancer de Montpellier - Val d'Aurelle (Other); Ente Ospedaliero Cantonale, Ticino, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 6363
Record Dates: First submitted 2024-03-19; First posted 2024-03-26 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Ovary Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Retrospective cohort: Patients affected by High Grade Seruous Ovarian Cancer with mesenteric infiltration confirmed by diagnostic laparoscopy, from January 2021 to December 2023
  Interventions: Diagnostic Test: Computed Tomography
- Prospective cohort: Patients affected by High Grade Seruous Ovarian Cancer with mesenteric infiltration confirmed by diagnostic laparoscopy
  Interventions: Diagnostic Test: Computed Tomography

INTERVENTIONS:
Diagnostic Test: Computed Tomography — Computed Tomography done according to Clinical Practice to assess mesenteric involvment

SUMMARY:
To evaluate if CT features at diagnosis in patients with HGSOC can be used to build an Artificial Intelligence model capable of discerning the pathological involvement of the mesentery, assessing the potential impediments for an optimal debulking surgery and predicting the development of resistance to platinum based chemotherapeutic agents.

ELIGIBILITY:
Inclusion Criteria:

1. Women with confirmed HGSOC wiht mesenteric involvment
2. Age > 18 years
3. FIGO STAGE IIIB-IV
4. Primary diagnosis
5. Signed informed consent

Exclusion Criteria:

1. Non-serous high grade epithelial ovarian cancer (serous low grade, mucinous, clear cell carcinoma, endometrioid or non-epithelial ovarian cancer)
2. Early stage disease (I and II stage)
3. CT scan not available
4. Non-primary diagnosis or patient subjected to neoadjuvant chemotherapy

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Women with confirmed HGSOC who exhibited mesenteric disease, including mesenteric retraction or diffuse mesenteric carcinomatosis, during diagnostic laparoscopy (or without mesenteric disease for the control cohort)
Sampling Method: Non-Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Preoperative Artificial Intelligence assisted CT-based evaluation | 1 year
  Preoperative Artificial Intelligence assisted CT-based prediction of patients with suboptimal debulking at surgery due to diffuse mesenteric disease or mesenteric retraction.

SECONDARY OUTCOMES:
Evaluation of the Radiologist Assessment of the CT | 1 year
  Identification of mesenteric infiltration from CT images using Artificial Intelligence at a comparable performance with human/radiologist assessment.
Prediction of Platinum Resistance | 1 year
  AI-assisted CT-based prediction of patients who will develop platinum resistance
Prediction of Progression Free Survival (PFS) and Overall Survival (OS) | 2 years
  Prediction of Progression Free Survival (PFS) and Overall Survival (OS) with Artificial Intelligence

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Panico, Dr, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Advanced Radiology Center, Roma, Italy

IPD SHARING:
Plan to Share IPD: No